CLINICAL TRIAL: NCT03672123
Title: GDF-15 Levels in Risk Stratification in Acute Pulmonary Embolism
Status: Completed | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Collaborators: National Science Center, Poland (Unknown)
Responsible Party: Principal Investigator, Marta Skowronska, Principal Investigator, Medical Doctor, Medical University of Warsaw
Other Study IDs: GDF-15 APE
Record Dates: First submitted 2018-09-05; First posted 2018-09-14 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Pulmonary Embolism
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum/plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- APE with RVD: RVD (right ventricle disfunction) defined according to ESC (European Society of Cardiology) criteria
- APE without RVD: RVD defined according to ESC criteria

SUMMARY:
Prospective observational study evaluating serum GDF-15 levels in patients with acute pulmonary embolism.

DETAILED DESCRIPTION:
Prospective observational study evaluating serum GDF-15 levels in patients with acute pulmonary embolism (APE).

In APE right ventricle failure developing due to ischemia and myocarditis is considered the primary cause of death, however, its pathomechanism has not been fully established yet. Growth differentiation factor 15 (GDF-15) is a chemokine secreted by activated macrophages in response to oxidative stress. It has now been shown that ischemic injury, mechanical stretch, and pro-inflammatory cytokines also stimulate the expression of GDF-15 in cardiac myocytes. The objective of this project is to describe the role of GDF-15 in the pathomechanism of acute right ventricle failure in the setting of acute pulmonary embolism and to verify the hypothesis that higher serum concentrations of GDF-15 are associated with more advanced right ventricle dysfunction and failure.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with APE hospitalized who give written consent.

Exclusion Criteria:

* lack of informed consent
* APE with symptoms lasting above 14 days before the admission
* acute coronary syndrome, diagnosed pulmonary hypertension
* severe valve disease
* sepsis
* active malignancy
* diagnosed mitochondrial diseases
* chronic kidney disease at least stage 4 (KDIGO)
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit 270 patients.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
hemodynamic deterioration | assessed daily through study completion, average of 10 days
  Hemodynamic deterioration defined according to ESC criteria as:
  change in blood pressure defined as: drop in systolic arterial blood pressure < 90 mmHg or at least 40 mmHg, lasting ≤ than 15 minutes

SECONDARY OUTCOMES:
Hemorrhagic complications | assessed daily through study completion, average of 10 days
  Major bleeding defined according to ISTH (International Society on Thrombosis and Haemostasis) criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Z Skowronska, MD, Principal Investigator — Medical University of Warsaw; Piotr Pruszczyk, Prof., Study Director — Medical University of Warsaw
Locations (1):
- Department of Internal Medicine & Cardiology with the Centre for Management of Venous Thromboembolic Disease, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No